CLINICAL TRIAL: NCT01087385
Title: Troponin T as Risk Stratification Tool in Patients With Peripheral Arterial Occlusive Disease
Brief Title: Troponin T as Risk Stratification Tool in Peripheral Arterial Occlusive Disease
Status: Completed | Type: Observational
Sponsor: University Heart Center Freiburg - Bad Krozingen (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Birgit Linnemann, Dr. Birgit Linnemann, University Heart Center Freiburg - Bad Krozingen
Other Study IDs: EK-Nr. 59/10
Record Dates: First submitted 2010-03-15; First posted 2010-03-16 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Peripheral Arterial Occlusive Disease
Keywords: peripheral arterial occlusive disease; mortality; cardiovascular events; amputation; peripheral arterial revascularization
MeSH Terms: conditions — Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Troponin T elevation
- No troponin T elevation

SUMMARY:
Study hypothesis: elevated Troponin T is a marker of increased mortality in patients with peripheral arterial occlusive disease (PAOD).

DETAILED DESCRIPTION:
Troponin T and I are established risk markers in patients with acute coronary syndrome. Only recently, troponin I was found to be elevated in patients with acute critical limb ischaemia. In another study, troponin I was associated with a higher mortality in patients with chronic critical limb ischaemia followed over two years. In a longitudinal study design we intend to follow all patients that were treated for symptomatic PAOD (Fontaine stages II-IV) from 01/2007 to 12/2007 in our department of angiology. Main outcome parameters are death and the occurrence of major vascular events and revascularization procedures during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic peripheral arterial occlusive disease
* aged >/= 18 years

Exclusion Criteria:

* unstable angina or acute coronary syndrome < 14 days
* percutaneous coronary intervention < 14 days
* other interventions or disease associated with troponin T release (i.e., acute pulmonary embolism, aortic dissection, heart valve replacement, acute heart failure, non-ischemic cardiomyopathy, heart surgery, thoracic trauma, endocarditis, myocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with peripheral arterial occlusive disease (Fontaine stages II-IV)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Death | 1 year

SECONDARY OUTCOMES:
Myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, stroke, amputation, peripheral revascularization, target limb revascularization, target vessel revascularization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Linnemann, M.D., Principal Investigator — Heart Center Bad Krozingen, Germany
Locations (1):
- Angiologie, Herzzentrum Bad Krozingen, Bad Krozingen, Germany

REFERENCES:
- [Derived] Linnemann B, Sutter T, Herrmann E, Sixt S, Rastan A, Schwarzwaelder U, Noory E, Buergelin K, Beschorner U, Zeller T. Elevated cardiac troponin T is associated with higher mortality and amputation rates in patients with peripheral arterial disease. J Am Coll Cardiol. 2014 Apr 22;63(15):1529-38. doi: 10.1016/j.jacc.2013.05.059. Epub 2013 Jun 21. PMID 23792625
- [Derived] Linnemann B, Sutter T, Sixt S, Rastan A, Schwarzwaelder U, Noory E, Buergelin K, Beschorner U, Zeller T. Elevated cardiac troponin T contributes to prediction of worse in-hospital outcomes after endovascular therapy for acute limb ischemia. J Vasc Surg. 2012 Mar;55(3):721-9. doi: 10.1016/j.jvs.2011.10.024. Epub 2012 Jan 24. PMID 22277685